CLINICAL TRIAL: NCT02900248
Title: Patients Diagnosed With Advanced Malignancy or Myelodysplasia, Tested by Standardized Sequencing, and Treated by Physician-Determined Care Plan: A CureOne Observational Registry (N1)
Brief Title: CureOne Registry: Advanced Malignancy or Myelodysplasia, Tested by Standard Sequencing and Treated by Physician Choice
Acronym: N1
Status: Terminated | Type: Observational
Why Stopped: Registry was built to handle Medicare coverage decision on NGS, but CMS decided to not require data.
Sponsor: CureOne (Other)
Responsible Party: Sponsor
Other Study IDs: N1OR
Record Dates: First submitted 2015-06-18; First posted 2016-09-14 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms; Lung Neoplasms; Colon Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Prostate Neoplasms; Kidney Neoplasms; Liver Neoplasms; Rectal Neoplasms; Hematologic Neoplasms; Multiple Myeloma; Myelodysplastic Syndromes; Ovarian Neoplasms; Bladder Neoplasms; Testicular Neoplasms; Endometrial Neoplasms; Brain Neoplasms; Biliary Tract Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Skin Neoplasms; Melanoma; Gastric Neoplasms; Anal Neoplasms; Sarcoma
Keywords: Biomarkers; High-Throughput Nucleotide Sequencing; Neoplasms; Myelodysplastic Syndromes
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Colonic Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Liver Neoplasms; Rectal Neoplasms; Hematologic Neoplasms; Multiple Myeloma; Myelodysplastic Syndromes; Ovarian Neoplasms; Urinary Bladder Neoplasms; Testicular Neoplasms; Endometrial Neoplasms; Brain Neoplasms; Biliary Tract Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Skin Neoplasms; Melanoma; Stomach Neoplasms; Anus Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Provider Determined Treatment: Participants with advanced solid or hematologic malignancy or myelodysplasia (MDS), will have their tumor or tissue tested by a standardized next generation sequencing (NGS) panel. They will be treated by physician determined treatment including FDA approved or compendia-listed biomarker directed therapy. All patients will be followed for time to progression by line of therapy, overall survival by line of therapy.
  Interventions: Other: Provider determined

INTERVENTIONS:
Other: Provider determined — Provider will treat patient as he/she feels best

SUMMARY:
Registry participants with advanced malignancy or myelodysplasia will have a sample of their tumor or tissue analysed for genetic alterations using next generation sequencing (NGS) performed in a lab that has been certified to meet a high quality standard. Treatments and outcomes will be reported to the registry to allow further understanding of how genetic differences can lead to better diagnosis and treatments.

DETAILED DESCRIPTION:
Every malignancy or myelodysplasia is different on a molecular (genetic) level even in patients with the same diagnosis. These differences often give prognostic information, determine what types of treatments are available for a patient, as well as determine outcomes. In this registry, the method of identifying the genetic difference of the disease (using Next Generation Sequencing or NGS) is standardized, the treatments received by a patient, and the outcome of these treatments are entered into a database where all identifying information is removed.

Payers (insurance companies) or others will generally pay for the testing, laboratories will report the genetic information, physicians and eventually patients will report treatments and outcomes. This information will then be reviewed frequently and analyzed to find better methods to improve the testing or treatments of disease.

It is expected that dozens of other trials or registries will eventually be available for participants.

ELIGIBILITY:
Inclusion:

1. Patient is ≥ 18 years old.
2. Patient is able to understand and agrees to comply with the requirements of the study and provides written informed consent indicating voluntary consent to participate in the registry. If the patient is unable to provide consent, but is able to comply with other study requirements, informed consent must be obtained by a durable power of attorney or healthcare proxy.
3. Patient is diagnosed with any of the following malignancies or disorders AND with the corresponding American Joint Commission on Cancer (AJCC) 7th Edition Staging OR listed clinical scenario (i.e. a patient initially diagnosed with early stage lung cancer would not be a candidate, but if they later developed metastatic disease, they would be eligible and could be enrolled in this registry):

   1. Solid Malignancies Tumor Type (Initial Stage: Clinical Scenario) Lung and Bronchus (Stage IIIB or IV: Metastatic or Extensive) Colorectal (Stage IVB: Metastatic) Pancreas (Stage IV: Metastatic) Breast (Stage IV: Metastatic) Prostate (Stage IV: Castrate resistant) Hepatobiliary (Non-resectable: Metastatic) Tumor of Unknown Primary (Non-resectable: Initial Diagnosis) Bladder (Stage IV: Metastatic) Esophageal (Stage IV: Metastatic) Brain and CNS (All: Initial Diagnosis) Ovarian Cancer (Stage IV or Non-resectable: Recurrent) Kidney or Renal Pelvis (Stage IV: Metastatic) Stomach (Stage IV: Metastatic) Endometrial (Stage IV: Metastatic) Melanoma (Stage IV: Metastatic) Oral Cavity and Pharynx (Stage IVC: Metastatic) Less common Solid Malignancies* (Stage IV: Metastatic)

      *Defined as <1% annual death rate in the SEER database. This also includes histologies of common tumors that have been shown to have a more aggressive phenotype and require a different treatment approach than their more common counterparts.
   2. Hematologic Malignancies Tumor Type (Initial Stage: Clinical Scenario) Non-Hodgkins Lymphoma (N/A: Progressed or relapsed after initial treatment) Multiple Myeloma (Non-smoldering disease: Requiring Treatment) Acute Myelogenous Leukemia (N/A: Initial Diagnosis or Relapse) Chronic Lymphocytic Leukemia (N/A: Progressed or relapsed after initial therapy) Acute Lymphoblastic Leukemia (N/A: Initial Diagnosis or Relapse) Hodgkins Lymphoma (N/A: Progressed or relapsed after initial therapy) Chronic Myelogenous Leukemia (N/A: Progressed or relapsed after initial therapy) Less common Hematologic Malignancies (N/A: Requiring Treatment)
   3. Myelodysplasia with cytopenias at time of requiring treatment
4. Unless otherwise specified, all participants will have NGS testing of an appropriate somatic tissue specimen (biopsy tissue or cell-free DNA) at a CureOne approved lab using the testing outlined in the protocol. The specimen used for testing must have been obtained within 6 months (180 days) preceding consent or on a specimen(s) obtained within 3 months (90 days) following consent to participate in this observational registry. Any non-registry biomarker testing must also be reported. Patient will be treated by physician-determined care plan.
5. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at initial screening.
6. Patient is willing and able to be treated by physician-determined care plan.
7. Patient may participate in other clinical studies or registries while participating in this observational registry.
8. Patient agrees with regular follow up (see Assessment Schedule below).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced malignancy or myelodysplasia
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Best Overall Response | 5 years
  Best overall response by line of therapy and biomarker
Time to Treatment Progression | 5 years
  Physician-determined Time to Treatment Progression by line of therapy and method of determining progression (worsening of disease, new lesions, clinical decline, and/or other).

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall survival by biomarker
Establish stable estimates of biomarker prevalence in patients with advanced malignancies in a large population. | 5 years
  Establish stable estimates of biomarker prevalence in patients with advanced malignancies in a large population.
To determine rate of enrollment into existing and future therapeutic clinical trials. | 5 years
  To determine rate of enrollment into existing and future therapeutic clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, M.D., Principal Investigator — Moores Cancer Center, University of California at San Diego; John Pfeifer, M.D., Ph.D., Study Chair — Washington University School of Medicine; Dane J. Dickson, M.D., Study Director — CureOne/Knight Cancer Center, Oregon Health and Science University
Locations (1):
- Teton Cancer Institute, Idaho Falls, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genomic and general outcome information will be available for further research through curated independent research projects

REFERENCES:
- [Background] Herbst RS, Prager D, Hermann R, Fehrenbacher L, Johnson BE, Sandler A, Kris MG, Tran HT, Klein P, Li X, Ramies D, Johnson DH, Miller VA; TRIBUTE Investigator Group. TRIBUTE: a phase III trial of erlotinib hydrochloride (OSI-774) combined with carboplatin and paclitaxel chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5892-9. doi: 10.1200/JCO.2005.02.840. Epub 2005 Jul 25. PMID 16043829
- [Background] Yang JC, Sequist LV, Geater SL, Tsai CM, Mok TS, Schuler M, Yamamoto N, Yu CJ, Ou SH, Zhou C, Massey D, Zazulina V, Wu YL. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2, LUX-Lung 3, and LUX-Lung 6. Lancet Oncol. 2015 Jul;16(7):830-8. doi: 10.1016/S1470-2045(15)00026-1. Epub 2015 Jun 4. PMID 26051236
- [Background] Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, Li W, Hou M, Shi JH, Lee KY, Xu CR, Massey D, Kim M, Shi Y, Geater SL. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Feb;15(2):213-22. doi: 10.1016/S1470-2045(13)70604-1. Epub 2014 Jan 15. PMID 24439929
- [Background] Peters S, Michielin O, Zimmermann S. Dramatic response induced by vemurafenib in a BRAF V600E-mutated lung adenocarcinoma. J Clin Oncol. 2013 Jul 10;31(20):e341-4. doi: 10.1200/JCO.2012.47.6143. Epub 2013 Jun 3. No abstract available. PMID 23733758
- [Background] Kohno T, Nakaoku T, Tsuta K, Tsuchihara K, Matsumoto S, Yoh K, Goto K. Beyond ALK-RET, ROS1 and other oncogene fusions in lung cancer. Transl Lung Cancer Res. 2015 Apr;4(2):156-64. doi: 10.3978/j.issn.2218-6751.2014.11.11. PMID 25870798
- [Background] Drilon A, Wang L, Arcila ME, Balasubramanian S, Greenbowe JR, Ross JS, Stephens P, Lipson D, Miller VA, Kris MG, Ladanyi M, Rizvi NA. Broad, Hybrid Capture-Based Next-Generation Sequencing Identifies Actionable Genomic Alterations in Lung Adenocarcinomas Otherwise Negative for Such Alterations by Other Genomic Testing Approaches. Clin Cancer Res. 2015 Aug 15;21(16):3631-9. doi: 10.1158/1078-0432.CCR-14-2683. Epub 2015 Jan 7. PMID 25567908
- [Background] Boland JF, Chung CC, Roberson D, Mitchell J, Zhang X, Im KM, He J, Chanock SJ, Yeager M, Dean M. The new sequencer on the block: comparison of Life Technology's Proton sequencer to an Illumina HiSeq for whole-exome sequencing. Hum Genet. 2013 Oct;132(10):1153-63. doi: 10.1007/s00439-013-1321-4. Epub 2013 Jun 12. PMID 23757002
- [Background] Jones S, Anagnostou V, Lytle K, Parpart-Li S, Nesselbush M, Riley DR, Shukla M, Chesnick B, Kadan M, Papp E, Galens KG, Murphy D, Zhang T, Kann L, Sausen M, Angiuoli SV, Diaz LA Jr, Velculescu VE. Personalized genomic analyses for cancer mutation discovery and interpretation. Sci Transl Med. 2015 Apr 15;7(283):283ra53. doi: 10.1126/scitranslmed.aaa7161. PMID 25877891
- [Background] Cappuzzo F, Bemis L, Varella-Garcia M. HER2 mutation and response to trastuzumab therapy in non-small-cell lung cancer. N Engl J Med. 2006 Jun 15;354(24):2619-21. doi: 10.1056/NEJMc060020. No abstract available. PMID 16775247
- [Background] Falchook GS, Janku F, Tsao AS, Bastida CC, Stewart DJ, Kurzrock R. Non-small-cell lung cancer with HER2 exon 20 mutation: regression with dual HER2 inhibition and anti-VEGF combination treatment. J Thorac Oncol. 2013 Feb;8(2):e19-20. doi: 10.1097/JTO.0b013e31827ce38e. No abstract available. PMID 23328556
- [Background] Cappuzzo F, Ligorio C, Toschi L, Rossi E, Trisolini R, Paioli D, Magrini E, Finocchiaro G, Bartolini S, Cancellieri A, Hirsch FR, Crino L, Varella-Garcia M. EGFR and HER2 gene copy number and response to first-line chemotherapy in patients with advanced non-small cell lung cancer (NSCLC). J Thorac Oncol. 2007 May;2(5):423-9. doi: 10.1097/01.JTO.0000268676.79872.9b. PMID 17473658
- [Background] Ou SH, Kwak EL, Siwak-Tapp C, Dy J, Bergethon K, Clark JW, Camidge DR, Solomon BJ, Maki RG, Bang YJ, Kim DW, Christensen J, Tan W, Wilner KD, Salgia R, Iafrate AJ. Activity of crizotinib (PF02341066), a dual mesenchymal-epithelial transition (MET) and anaplastic lymphoma kinase (ALK) inhibitor, in a non-small cell lung cancer patient with de novo MET amplification. J Thorac Oncol. 2011 May;6(5):942-6. doi: 10.1097/JTO.0b013e31821528d3. PMID 21623265
- [Background] Drilon A, Wang L, Hasanovic A, Suehara Y, Lipson D, Stephens P, Ross J, Miller V, Ginsberg M, Zakowski MF, Kris MG, Ladanyi M, Rizvi N. Response to Cabozantinib in patients with RET fusion-positive lung adenocarcinomas. Cancer Discov. 2013 Jun;3(6):630-5. doi: 10.1158/2159-8290.CD-13-0035. Epub 2013 Mar 26. PMID 23533264
- [Background] Falchook GS, Ordonez NG, Bastida CC, Stephens PJ, Miller VA, Gaido L, Jackson T, Karp DD. Effect of the RET Inhibitor Vandetanib in a Patient With RET Fusion-Positive Metastatic Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 May 20;34(15):e141-4. doi: 10.1200/JCO.2013.50.5016. Epub 2014 Nov 3. No abstract available. PMID 25366691
- [Background] Shaw AT, Ou SH, Bang YJ, Camidge DR, Solomon BJ, Salgia R, Riely GJ, Varella-Garcia M, Shapiro GI, Costa DB, Doebele RC, Le LP, Zheng Z, Tan W, Stephenson P, Shreeve SM, Tye LM, Christensen JG, Wilner KD, Clark JW, Iafrate AJ. Crizotinib in ROS1-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Nov 20;371(21):1963-71. doi: 10.1056/NEJMoa1406766. Epub 2014 Sep 27. PMID 25264305